CLINICAL TRIAL: NCT06487026
Title: An Extension Study to Evaluate the Safety of ArcBlate MRgHIFU in Patients With Painful Bone Metastases
Brief Title: Safety of ArcBlate MRgHIFU in Patients With Painful Bone Metastases: An Extension Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: EpiSonica (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTP-BM-23-01
Record Dates: First submitted 2024-06-27; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-06

CONDITIONS: Bone Metastases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRgHIFU treatment arm (Experimental): Subjects will receive MRgHIFU treatment by using ArcBlate Focused Ultrasound Ablation System.
  Interventions: Device: ArcBlate Focused Ultrasound Ablation System

INTERVENTIONS:
Device: ArcBlate Focused Ultrasound Ablation System — MR-guided High Intensity Focused Ultrasound (MRgHIFU)

SUMMARY:
An Extension Study to Evaluate the Safety of ArcBlate MRgHIFU in Patients with Painful Bone Metastases

DETAILED DESCRIPTION:
Pain palliation of bone metastasis through localized denervation by thermal ablation.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, who randomized into Sham control group and withdrew from CTP-BM-22-01 Study (i.e. main study) due to lack of efficacy.
2. Completed 14-day evaluation in main study.
3. Will provide completed and signed written informed consents.

Exclusion Criteria:

1. Pregnant women.
2. Subjects who do not meet any of the inclusion criteria in CTP-BM-22-01 Study (i.e. main study) after re-evaluation.
3. Determined by the investigator to be not suitable for the conduct of the study for any other reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Unanticipated adverse device effects (UADEs) from Day 0 to 90. | from Day 0 to 90
  UADEs is defined as any serious adverse effect on health or safety or any life-threatening problem or death caused by, or associated with, a device, if that effect, problem, or death was not previously identified in nature, severity, or degree of incidence in the investigational plan or application (including a supplementary plan or application), or any other unanticipated serious problem associated with a device that relates to the rights, safety, or welfare of subjects.

SECONDARY OUTCOMES:
Solicited events from Day 0 to 30 | from Day 0 to 30
  Major adverse events (Day 0 to 7)、Solicited adverse events (Day 0 to 30)
Unsolicited adverse events from Day 0 to 90 | from Day 0 to 90
  Unsolicited adverse events are defined as whose nature or intensity are not consistent with the solicited AE.

CONTACTS AND LOCATIONS:
Locations (4):
- Taiwan (4):
  - Far Eastern Memorial Hospital, New Taipei City
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Chang Gung Memorial Hospital - Linkou, Taoyuan District

IPD SHARING:
Plan to Share IPD: No